CLINICAL TRIAL: NCT03901547
Title: An Education and Behavioral, Single-center, Observational Cohort Study Evaluating the Effect of Emotion Regulation and Burnout on Medical Trainees' Learning and Documentation of Serious Illness Communication
Brief Title: Emotion Regulation and Burnout Impact on Communication Documentation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Combination of no funding and time commitments on PI
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Garrett T. Wasp, Fellow, GME Hematology-Oncology, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: D19033
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Communication
Keywords: documentation; serious illness
MeSH Terms: conditions — Communication | interventions — Maslach Burnout Inventory

STUDY DESIGN:
Intervention Model Description: Both groups get the same education intervention. Tier two gets additional measurement intervention and one additional system based intervention (e.g. priming) that Tier 1 does not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education and Documentation (Tier 1) (Other): Education only. Participants who do not wish to enroll in the behavioral observation group are followed in the education only. This includes participation in a two week palliative medicine elective which is a part of the medical trainees training and training in the serious illness communication guide (SICG). Participants can opt out of the pre and post training confidence surveys, and simulated patient encounters. Electronic documentation of the SICG by these trainees will be monitored prospectively. Participants will be provided reminders and profile information on their own documentation rate of the SICG via email and have the ability to opt out of receiving emails if they wish.
  Interventions: Behavioral: Communication Skills Training; Behavioral: Profile feedback
- Priming and additional measures (Tier 2) (Other): Education and behavioral observation cohort. These participants must sign an informed consent to participate in this part of the study. In addition to all of Tier 1 activities, participants also complete psychological inventories at three time points to measure emotion regulation and burnout, and participate in a semi-structured interview.
  Interventions: Behavioral: Communication Skills Training; Behavioral: Profile feedback; Other: Maslach burnout inventory; Other: Emotion Regulation Skills Question (ERSQ); Other: Semi-structured interview; Behavioral: Priming

INTERVENTIONS:
Behavioral: Communication Skills Training — Education training in the serious illness communication guide (SICG) by Ariadne labs.
Behavioral: Profile feedback — Providing participants their personal documentation rate of SICG in the electronic medical record
Other: Maslach burnout inventory — Maslach burnout inventory
  Arms: Priming and additional measures (Tier 2)
Other: Emotion Regulation Skills Question (ERSQ) — This validated instrument consists of 27 items, and includes subscales related to nine competencies of coping with negative emotion (awareness, sensations, clarity, understanding, acceptance, tolerance, readiness to confront, compassionate self-support and modification) which can be summed to a total score (TOTAL). This validated instrument consists of 27 items, and includes subscales related to nine competencies of coping with negative emotion (awareness, sensations, clarity, understanding, acceptance, tolerance, readiness to confront, compassionate self-support and modification) which can be summed to a total score (TOTAL).
  Arms: Priming and additional measures (Tier 2)
Other: Semi-structured interview — Interviewer asked subjects are a series of questions based on interview guide. Current guide designed to assess subject perception of implementation of training in clinical encounters, most recent encounter with patient with serious illness, barriers to documentation and coaching by faculty on communication. Interviews will be recorded and expected duration is 20-40 minutes.
  Arms: Priming and additional measures (Tier 2)
Behavioral: Priming — Participants will be provided a list of 30 patients they have encountered before that 1) have at least one documented note and 2) have a high probability for having serious illness as determined by electronic medical record screening. Participants will be asked 4 "yes or no" questions on each patient. Questions: 1) do you believe this patient has serious illness?; 2) would you be surprised if this patient died in the next year?; 3) would the patient benefit from the serious illness conversation guide? and 4) If you saw this patient again, would you use the serious illness conversation guide with him/ her?
  Arms: Priming and additional measures (Tier 2)

SUMMARY:
This is a single-institution cohort study with two tiers. All participants receive the interventions in Tier 1. Tier 1 is an education study where participants can complete electronic surveys on their pre and post intervention confidence, perform two simulated patient encounters and have their documentation of electronic template monitored longitudinally over 12 months. Participants are free to opt out of any activity related to education assessment or system-based interventions to promote the use of learned skills (e.g. priming or profile feedback). Signed informed consent will Not be required for this tier. Tier 2 includes additional measurements to the Tier 1 activities, and a priming intervention (e.g. provided the names of patients they have have). Participants in Tier 2 complete psychological inventories at three time points to measure emotion regulation and burnout, and participate in a semi-structured interview. after completing the training, they will complete a "priming" intervention. The investigators will require signed informed consent to participate in Tier 2.

DETAILED DESCRIPTION:
Before Communication Training Activities Tier 1 (education-only subjects): Three to four weeks prior to the subject's two-week palliative care elective they will be sent an email to complete an online confidence survey. They will receive email reminders to complete the survey until survey is completed.

Tier 2 (education + psychological measurements of subjects): Subjects will have reviewed and signed consent documentation. In addition to the above online confidence survey, they will also receive email to complete electronic ERSQ and MBI.

Two week palliative care elective Tier 1 - Integrated into the two-week elective with the palliative care department, subjects undergo a 1) four-hour training focused on the SICG©; 2) two simulated patient encounters with trained actors and feedback provided after training, 3) participant sent electronic notification to take post intervention survey of confidence Tier 2 - In addition to above, these subjects will also complete a Priming intervention. They will receive a list of patients whom 1) the study subjected documented at least one note on in the past and 2) have a high likelihood of serious illness as determined by an electronic process. This list will be shared securely through Dartmouth secure file electronically, and participants will be asked four "yes or no" questions for each patient: 1) do they believe the patient has serious illness?; 2) would you be surprised if the patient died within the next year?, 3) Is this patient an appropriate patient to use the serious illness conversation guide? and 4) If you saw this patient again, would you use the serious illness conversation guide with him/ her? Subjects will be asked to review no more than 30 patients. Subjects will be asked to return the completed email via Dartmouth secure file share.

Electronic communication every two months following completion of elective Tier 1 - Every two months after completing the training, participants will receive email compare his or her own documentation of the taught template to top and average performers (comparison results given are anonymous). Non-top and top performers will receive different messages, customized through pre-testing with non-study residents and fellows. For example: "Talking to patients about their values is important but can take some pre-visit planning. Choose a patient you will see in the next two weeks to use the SICG" (non top-performers) or "Good job! Talking to patients about their values is important. The way we continue to improve is by having more conversations. Choose a patient you will see in the next two weeks to use the SICG." (top-performers). At four months, subjects will be asked electronically to complete their final confidence survey.

Tier 2 - For this part of the study, identical to Tier 1

Semi-structured interviews Tier 2 only - Planned to occur about three months following training. Subjects are asked a series of questions designed to assess subject perception of serious illness communication, obstacles to implementing the training in practice, barriers to documentation and coaching sessions in real patient encounters with trained faculty. Interviews will be recorded, and expected duration is 20-40 minutes.

Simulated Patient encounter at six months Tier 1 - Subject is contacted to arrange one-hour for simulated patient encounter, about 20-30 minutes for skill practice and the remainder for debrief. Subject has permission from program to have this hour to be away from their clinical duties.

Tier 2 - identical to Tier 1.

Six and 12 month ERSQ and MBI assessment Tier 2 only - emails will be sent to subject to take ERSQ and MBI at month six and 12 following training

ELIGIBILITY:
Inclusion Criteria:

* All second year (PGY-2) internal medicine residents
* All hematology-oncology fellows

Exclusion Criteria:

* Missed more than five days of the palliative care education elective

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Template use at 12 months | 12 months following training
  Documentation events in the electronic medical record using the dot-phrase or electronic template for the serious illness conversation guide

SECONDARY OUTCOMES:
post-intervention self-rated confidence | Pre intervention and 4 months post intervention
  Using a 5 point Likert scale (i.e. 1=strongly disagree, 2=disagree, 3=neutral, 4=agree 5=strongly agree) participants were asked to rate their confidence in various communication skills domains pre- and post-intervention via online survey. The current version has 12 items that trainees rate their post-intervention confidence
performance in simulated patient encounters | Intervention start, 2 weeks and 6 months
  Performance is measured by an internally developed checklist. A single independent observer, during simulated patient encounters, will evaluate trainees. One point is assigned for each item used by the trainee. The checklist contains three scores: conversation guide specific items (16 points), global communication skills (9 points), and a combined score (25 points). This checklist was developed internally and based on the experience training residents in the Serious Illness Conversation Guide (SICG).
semi-structured interview responses | 4 months
  Interviewer uses a semi-structured interview guide to ask open ended questions to participants. The current verison of the interview guide assesses participant experience in 3 broad areas: experience using training in clinical practice, most recent encounter with a patient with serious illness and experience receiving faculty coaching in communication skills. Interviews generally range from 15 to 40 minutes in length. Conversations will be recorded, transcribed, and analyzed qualitative for theme and content.
emotion regulation skills | start, 6 months and 12 months
  The emotion regulation skills questionnaire (ERSQ) is a validated instrument consists of 27 items, and includes subscales related to nine competencies of coping with negative emotion (awareness, sensations, clarity, understanding, acceptance, tolerance, readiness to confront, compassionate self-support and modification) which can be summed to a total score (TOTAL). The ERSQ assesses each skill by means of three items introduced by the phrase "In the last week…" and answered on a 5-point Likert-scale. Higher scores indicate stronger emotion regulation skills. The investigators will administer the ERSQ via online survey
Change in Burnout | Baseline, 6 months and 12 months
  The responses to the Maslach Burnout Inventory tool will be evaluated to measure change in burnout. This validated, psychological inventory consists of 22 items related to occupational burnout, and includes subscales related to Emotional exhaustion (EE; 9 items), Depersonalization (DP; 5-items), and Personal Accomplishment (PA; 8 items). The MBI assesses each item on a 7-point Likert-scale. Higher scores indicated greater burnout. The investigators will use the MBI / Human Services Survey for Medical Personnel administered via online survey

CONTACTS AND LOCATIONS:
Overall Officials: Garrett T Wasp, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
At this point no plans to share individual data outside of study team. If study data were to be shared, the investigators would need to make sure it was anonymous and could not be traced back to specific individuals inn order to protect our participants

REFERENCES:
- [Background] Bernacki R, Hutchings M, Vick J, Smith G, Paladino J, Lipsitz S, Gawande AA, Block SD. Development of the Serious Illness Care Program: a randomised controlled trial of a palliative care communication intervention. BMJ Open. 2015 Oct 6;5(10):e009032. doi: 10.1136/bmjopen-2015-009032. PMID 26443662
- [Background] Berking M, Poppe C, Luhmann M, Wupperman P, Jaggi V, Seifritz E. Is the association between various emotion-regulation skills and mental health mediated by the ability to modify emotions? Results from two cross-sectional studies. J Behav Ther Exp Psychiatry. 2012 Sep;43(3):931-7. doi: 10.1016/j.jbtep.2011.09.009. Epub 2011 Nov 27. PMID 22406495
- [Background] Ebert DD, Christ O, Berking M. Entwicklung und validierung eines fragebogens zur emotionsspezifischen selbsteinschätzung emotionaler kompetenzen (SEK-ES). Diagnostica. 2013;59(1):17-32. doi:10.1026/0012-1924/a000079.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03901547/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03901547/ICF_001.pdf